CLINICAL TRIAL: NCT06860048
Title: Randomized Controlled Trial of Arm Sleeve and Forearm Fatigue During Robotic Surgery
Brief Title: Trial of Arm Sleeve and Forearm Fatigue During Robotic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Sydney (Other Government)
Responsible Party: Principal Investigator, Shing Wong, Associate Professor, Prince of Wales Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/ETH02203
Record Dates: First submitted 2025-02-25; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm sleeve (Active Comparator): Randomised to wear arm sleeve on left or right
  Interventions: Device: Arm sleeve

INTERVENTIONS:
Device: Arm sleeve — Randomised to wear arm sleeve on left or right

SUMMARY:
The study objective was to investigate whether wearing a forearm compression sleeve during robotic surgery reduces muscle fatigue as measured objectively by a grip strength dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Robotic surgeon

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle fatigue | 2 hours after intervention
  Hand grip strength (muscle fatigue)was assessed at the beginning and at the two-hour mark during the robotic console component of the surgical case, using the Camry Electronic Handgrip Dynamometer (CAMRY model: SCACAM-EH101). The non-sleeve-wearing forearm acted as a control. During testing, the surgeon sat upright with the elbows flexed at right angles by the side of the body and hands in neutral positions (halfway between supination and pronation). The handle was pulled with maximum force for three seconds. The hand grip strength (measured in kg force) was recorded ten times for the dominant (right) and non-dominant (left) hands alternately.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on reasonable request